CLINICAL TRIAL: NCT07110519
Title: Positron Emission Tomography (PET) Contrast Agent Kinetics and Safety: [18F]-Fluoromannitol
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PAKMANN
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Healthy; Adult; Age 18-75 years; Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Healthy adult volunteers who meet the eligibility criteria of the study.
  The study will evaluate the safety of [18F]-fluoromannitol as a tracer in healthy adult humans. Information will also be collected on the movement of the tracer in the body which may assist with diagnosing infections.
  Interventions: Drug: [18F]-fluoromannitol

INTERVENTIONS:
Drug: [18F]-fluoromannitol — [18F]-fluoromannitol is an investigational, novel radiotracer for use with PET scan imaging to help detect disease or infection.

SUMMARY:
This is a Phase 0 interventional, non-therapeutic study investigating the biodistribution and safety of [18F]-fluoromannitol as a radiotracer (a substance used to help detect disease or infection) in Positron Emission Tomography (PET) scans.

The primary objective of this study is to generate safety data in healthy adult human volunteers. In the future, this tracer may help to determine if a medical problem is infectious in people who have Sickle Cell Disease, cancer or other conditions that impact the immune system, or with people who have joint implants.

Primary Objective

- Generate safety data, biodistribution and perform human organ dosimetry for [18F]- fluoromannitol as a novel PET tracer.

Participants will be recruited primarily from St. Jude Children's Research Hospital employees and SJLIFE participants, and from the broader Memphis community if needed.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety and movement throughout the body of 18F-FMtl in healthy adult volunteers. It will be conducted under an IND approved by the FDA. The IND is required as 18F-fMtl is not commercially available and has not been studied in humans.

The design for this phase 0 study will be a single-group prospective trial.

Primary intervention is the administration of intravenous [18F]-fluoromannitol as a radiotracer with subsequent PET scans. Associated interventions include collection of blood and urine samples, vital signs, and symptoms from participants.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers, 18-75 years of age.

* Female participants of childbearing age must not be lactating due to theoretical potential harm to the infant from exposure to radiation.
* Informed consent signed by participant according to the guidelines of the institutional review board.

Exclusion Criteria:

Initial Eligibility Exclusion Criteria (Entry to Screening Phase -

* Participant currently has a fever or other symptoms concerning for an active infection or is currently undergoing treatment for an active infection.
* Participant has been diagnosed and/or treated for a known or suspected bacterial infection within the past 60 days.
* Participant has known disease of the lung, liver, kidneys, gastrointestinal tract, bones/joints, or known immune suppression or autoimmune disease that is likely to have active inflammation (examples to exclude: Crohn's disease, COPD; example to i include: well controlled asthma)
* Participant has prosthetic or indwelling device(s) currently or has had one in the past 60 days.
* Participant is pregnant or breastfeeding.
* Use of drugs known to have interaction or be affected by mannitol within 60 days of enrollment.
* Participant has any condition that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol, including being unable to tolerate the PET scan procedures.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
* Participant is currently participating in another study subject to an IND.

Final Eligibility Exclusion Criteria (Entry to Study):

At the time of the Final Eligibility Determination (Imaging Study Visit 1):

* Participant no longer meets one or more of the Inclusion Criteria
* Participant now fails one or more of the Initial Eligibility Exclusion Criteria
* Estimated glomerular filtration rate is < 45 ml/minute/1.73m2
* Positive pregnancy test (females only)
* One or more of the results from laboratory (hematology, chemistries, inflammatory markers), vital signs, or ECG specified in the schedule of evaluations is outside the normal institutional range AND is clinically significant in the opinion of the investigator.

Re-screening will not be allowed unless the Investigator considers the cause of the initial screen failure to be of an acute and/or completely reversible nature.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety of [18F]fluoromannitol administration in up to 10 human subjects. | Baseline at study entry and within 4 days following PET/CT.
  Safety will be assessed by the number and percentage of patients with adverse events following [18F]fluoromannitol administration. Adverse events will be categorized by the FDA's Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials.
Evaluate the biodistribution of [18F]fluoromannitol in up to 10 human subjects. | Through study completion, with an average of 3 months post-PET/CT.
  Calculate the absorbed dose of [18F]fluoromannitol in normal organs.

CONTACTS AND LOCATIONS:
Overall Officials: Kiel Neumann, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols